CLINICAL TRIAL: NCT07086222
Title: A Phase 4, Randomized, Double-Blind, Placebo-Controlled, Post-Marketing Study to Evaluate the Efficacy and Safety of an Omicron JN.1 Subvariant SARS-CoV-2 rS Vaccine Adjuvanted With Matrix-M® in Adults 50 to < 65 Years of Age Without High Risk Conditions for Severe COVID-19
Brief Title: Efficacy and Safety of NVX-CoV2705
Acronym: COVID-19
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019nCoV-420
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: COVID-19; Sars-CoV-2 Infection
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Matrix-M

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NVX-CoV2705 (Experimental): a single intramuscular (IM) injection of NVX-CoV2705 on Day 0
  Interventions: Biological: NVX-CoV2705
- Placebo (Placebo Comparator): a single intramuscular (IM) injection of placebo (normal saline) on Day 0
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: NVX-CoV2705 — NVX-CoV2705 vaccine in a 0.5 mL injection volume at an antigenic dose of 5 µg with 50 µg Matrix-M adjuvant
  Other Names: Omicron JN.1 subvariant SARS-CoV-2 rS vaccine adjuvanted with Matrix-M
  Arms: NVX-CoV2705
Biological: Placebo — Placebo (normal saline) in a 0.5 mL injection volume.
  Arms: Placebo

SUMMARY:
This is a Phase 4, post-market US study, evaluating the efficacy and safety of a single dose of the NVX-CoV2705 Omicron JN.1 COVID-19 vaccine. Approximately 6,500 healthy adults aged 50 to under 65 will be randomized to receive either the vaccine or a placebo, with follow-up for 180 days.

DETAILED DESCRIPTION:
This is a Phase 4, multicenter, randomized, double-blind, placebo-controlled, post-marketing study to evaluate the efficacy and safety of a single dose of an Omicron JN.1 subvariant severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) recombinant (r) spike (S) protein nanoparticle vaccine (SARS-CoV-2 rS) adjuvanted with Matrix-M (NVX-CoV2705) in adults 50 to < 65 years of age who are not considered to be at high risk of severe coronavirus disease 2019 (COVID-19). This study will be conducted in the United States (US).

Approximately 6,500 participants will be randomized in a 1:1 ratio via block randomization to receive a single intramuscular (IM) injection of NVX-CoV2705 or placebo (normal saline) on Day 0 and remain on study for efficacy and safety data collection through Day 180/end of study (EoS).

ELIGIBILITY:
Inclusion Criteria:

* To be included in this study, each individual must satisfy all of the following criteria:

  1. Adults 50 to < 65 years of age at time of study vaccination (Day 0) who are not considered to be at high risk of severe COVID-19.
  2. Participants unvaccinated to SARS-CoV-2 or participants previously vaccinated with a COVID-19 vaccine ≥ 90 days prior to study vaccination.
  3. Participant or legally acceptable representative is willing and able to give informed consent prior to study enrollment and to comply with study procedures.
  4. Female participants of childbearing potential (defined as any participant who has experienced menarche and who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea ≥ 12 consecutive months]) must agree to be heterosexually inactive from at least 28 days prior to enrollment and through 90 days after vaccination OR agree to consistently use a medically acceptable method of contraception listed below from ≥ 28 days prior to enrollment and through 90 days after vaccination.

     1. Condoms (male or female) with spermicide (if acceptable in country)
     2. Diaphragm with spermicide
     3. Cervical cap with spermicide
     4. Intrauterine device
     5. Oral or patch contraceptives
     6. Norplant®, Depo-Provera®, or other in country regulatory approved contraceptive method that is designed to protect against pregnancy
     7. Abstinence, as a form of contraception, is acceptable if in line with the participant's lifestyle NOTE: Periodic abstinence (eg, calendar, ovulation, sympto-thermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
  5. Agrees not to participate in any research involving receipt of investigational products (drug/biologic/device), including other SARS-CoV-2 prevention or treatment trials, for the duration of the study.

Exclusion Criteria:

* If an individual meets any of the following criteria, he or she is ineligible for this study:

  1. Is considered to be at high risk of severe COVID-19 due to underlying medical conditions or risk factors that demonstrated a conclusive increase in risk for at least one severe COVID-19 outcome, as described by the Centers for Disease Control and Prevention (CDC) .
  2. Unstable acute illness at the time of vaccination.
  3. Participation at the time of study enrollment or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.
  4. Current participation in any other COVID-19 prevention clinical trial.
  5. Known history of COVID-19 infection within 90 days of study vaccination.
  6. Any known history of allergies to products contained in the investigational product in the participant's lifetime.
  7. Any known history of anaphylaxis to any prior vaccine in the participant's lifetime.
  8. Known history of myocarditis or pericarditis in the participant's lifetime.
  9. Chronic administration (defined as > 14 continuous days) of immunosuppressant, systemic glucocorticoids, or other immune-modifying drugs within 90 days prior to study vaccination (Day 0).

     NOTE: An immunosuppressant dose of glucocorticoid is defined as a systemic dose ≥ 10 mg of prednisone per day or equivalent. The use of topical, inhaled, or intranasal glucocorticoids is permitted. Topical tacrolimus and ocular cyclosporin are permitted.
  10. Received immunoglobulin or blood-derived products within 90 days prior to study vaccination (Day 0).
  11. Participants who are pregnant, or who plan to become pregnant within 90 days following study vaccination.
  12. Any other condition that, in the opinion of the investigator, would pose a health risk to the participant if enrolled or could interfere with evaluation of the study vaccine or interpretation of study results (including neurologic or psychiatric conditions likely to impair the quality of safety reporting).
  13. Study team member or immediate family member of any study team member (inclusive of Sponsor, clinical research organization [CRO], and study site personnel involved in the conduct or planning of the study).

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6500 (Estimated)
Dates: Start 2025-11-10 (Estimated); Primary Completion 2026-01-09 (Estimated); Study Completion 2026-07-09 (Estimated)

PRIMARY OUTCOMES:
First episode of PCR-positive symptomatic COVID 19 | Day 0 to Day 180
  First episode of PCR-positive symptomatic COVID 19 from Day 0 (post vaccination) through Day 180/EoS

SECONDARY OUTCOMES:
First episode of PCR-positive symptomatic COVID 19 | Day 42 to Day 180
  First episode of PCR-positive symptomatic COVID 19 through Day 180/EoS
Participants with Medically attended adverse events (MAAEs), Serious adverse event (SAEs) and Adverse event of special interest (AESIs) | Day 180
  Number of participants reported MAAEs attributable to study vaccine, SAEs, or AESIs through Day 180/EoS.